CLINICAL TRIAL: NCT04318574
Title: The Effects of a 6-week Balance, Agility, Strengthening Exercise (BASE) Class on Balance Performance, Self-Efficacy, and Fear of Falling in Cancer Survivors
Brief Title: The Effects of a 6-week Balance, Agility, Strengthening Exercise Class
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Karen Dobbin, Principal Investigator, Clinical Instructor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2019:470
Record Dates: First submitted 2020-03-17; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Neoplasms
Keywords: Cancer; Balance impairment; Self-efficacy; Fear of falling; Balance training
MeSH Terms: conditions — Neoplasms | interventions — Alkalies; Artifacts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Balance, Agility, Strengthening Exercise (BASE) class intervention - a 6-week exercise class to determine the change in balance performance, fear of falling and self-efficacy
  Interventions: Other: Balance, Agility, Strengthening Exercise (BASE) Class

INTERVENTIONS:
Other: Balance, Agility, Strengthening Exercise (BASE) Class — The BASE class will be conducted twice weekly for 1.5 hours each session over a 6-week period and will include a 10-minute warm-up, 30 minutes of static and dynamic balance exercises, 20 minutes of lower extremity strengthening exercises, and a 10-minute cool-down. There will be weekly falls prevention and mobility enhancement education provided during the class.

SUMMARY:
Cancer treatments can have a significant impact on a cancer survivor's function and independence, and these patients can have twice the incidence of falls than their cancer-free peers. Balance programs of varying lengths have shown to improve balance performance, increase self-efficacy and decrease fear of falling; however, there are limited intervention studies amongst cancer survivors, and none that examine the combination of balance performance, self-efficacy and fear of falling. It is believed that this study will show that a 6-week Balance, Agility, Strengthening Exercise (BASE) Class is a sufficient time frame to demonstrate a positive effect on balance performance, self-efficacy, and fear of failing in cancer survivors, and will add to the body of knowledge in this population.

DETAILED DESCRIPTION:
Objectives Given that this combination of outcomes have not been sufficiently measured in the cancer population, and most balance and agility training programs are 12 weeks or more in length, the objectives of this study is to determine the effects of a 6-week intervention, the Balance, Agility, Strengthening Exercise (BASE) Class, on the balance performance, self-efficacy, and the fear of falling in cancer survivors.

Methods This study is a 3 year exercise interventional study, with 20 participants per year. In year one of the study, 20 participants will be enrolled in a 6-week Balance, Agility, Strengthening Exercise (BASE) Class. The pre-program data collection will include: demographic data; initial intake examination utilizing standard physiotherapy assessment of range of motion, flexibility, and strength; use of validated balance performance tools; and validated self-report surveys for balance confidence, fear of falling, and quality of life. The participants will attend the BASE class twice weekly for 6-weeks. The post-program data collection is to include the same outcome measures.

Subsequent years will be an observational study of the same design, enrolling 20 participants in year 2 and 3 for a 6-week BASE class. A total of 60 participants will be recruited over 3 years providing adequate power to assess program efficacy. Based on the resources available, this study can only accommodate 20 participants per year and can only be conducted for a 6-week period each year of the study.

Participants and recruitment Posters and hand bills will be distributed and placed throughout CancerCare recruiting participants for the study (self-referral). In addition, hand bills will provided for oncologists, oncology nurses, and psychosocial clinicians to give to patients/potential participants within the clinical areas at CancerCare. After receiving the hand bill with the study description and information, potential participants can choose to phone or e-mail the PI to indicate their interest in the study. A phone interaction will take place between the PI and potential participant to determine if they meet the inclusion criteria. Once it is determined that they meet the inclusion criteria, an in-person meeting will be arranged and they will be provided with the study's objectives, risks and benefits, and the consent document. Time will be allowed for the potential participant to ask questions and to consider their enrollment in the study. After a thorough discussion and review of the documents, the potential participant will be asked to sign the consent form. If requested, a person will be allowed to take the consent form home for further consideration prior to signing.

Data collection Prior to the start of the BASE Class, an initial assessment will take place. This assessment will utilize standard physiotherapy assessment of range of motion, flexibility, and strength; use of validated balance performance tools; and validated self-report surveys for balance confidence, fear of falling, and quality of life.

Intervention:

The BASE class will run twice weekly for 1.5 hours each session over a 6-week period and will include a 10-minute warm-up, 30 minutes of static and dynamic balance exercises, 20 minutes of lower extremity strengthening exercises, and a 10-minute cool-down. There will be weekly falls prevention and mobility enhancement education provided during the class.

Statistical Analysis Pre-post paired comparisons will be conducted for each balance performance and self-reported questionnaire measure. A paired T-test or Wilcoxon signed ranks test will be performed according to the observed distributions.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling
* ambulatory
* diagnosed with hematological or solid cancer tumors (except brain tumors/brain metastases)
* age >18 years
* self-identified as experiencing impaired balance, and scoring less than 80% on the Activities-specific Balance Confidence Scale
* able to communicate in English

Exclusion Criteria:

* metastatic cancer
* those unable to provide informed consent
* those having previously received physiotherapy and exercise instruction from the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-06 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Balance Performance - miniBest | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  Mini-Balance Evaluation Systems Test is a 14-item balance scale covering a broad spectrum of performance tasks including dynamic body stability, transfers, gait, variation of support surfaces, and of visual conditions, obstacle negotiation, reactions to external forces and performance during dual-tasking.
Balance Performane - TUG | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  Timed Up and Go: a rise from a chair, 3-meter walk, turn and walk back to chair and sitting. Designed to measure mobility, balance, and locomotor performance; evaluates falls risk and basic functional mobility.
Balance Performance - Timed Unipedal Stance Test | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  A simple test for measuring static aspects of balance ability, measured in seconds with eyes open and eyes closed; useful when combined with other balance performance tests.
Balance Performance - 6-meter Gait Speed Test | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  A 6-meter walking test measured in meters/second; an indicator of walking ability, function, and mobility.
Balance Performance - Four Square Step Test | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  A timed measurement of stepping whilst changing direction to provide a measure of dynamic standing balance and mobility; stepping forwards, sideways, and backwards over obstacles in a specified sequence.

SECONDARY OUTCOMES:
Self-report ABC Scale | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  Activities-specific Balance Confidence Scale is a 16-item self-report questionnaire examining a person's confidence in a broad range of activities with various difficulties; to assess balance confidence in ambulatory community-dwelling older adults
Self-report MFES | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  Modified Fall Efficacy Scale International is a 15 question self-rated scale assessing a person's confidence in performing activities in the home, plus additional items related to outdoor activities.
self-report Fear of Falling | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  A 14 item scale that examines fear of falling and the effect it has on participation in various activities
Self-report Quality of Life FACT-G | 1-2 weeks prior to BASE Class, change from baseline 1-2 weeks post BASE Class
  Functional Assessment of Cancer Therapy - General is a 27-item self-report instrument that consists of 4 sub-scales: physical well-being, social well-being, emotional well-being, and functional well-being to measure quality of life for cancer patients.

IPD SHARING:
Plan to Share IPD: No